CLINICAL TRIAL: NCT05097911
Title: A Phase 1 Study of RNA Oligonucleotide, MTL-CEBPA, Atezolizumab and Bevacizumab in Patients With Advanced Hepatocellular Carcinoma Without Previous Systemic Therapy.
Brief Title: Phase I Study of RNA Oligonucleotide, MTL-CEBPA, Atezolizumab and Bevacizumab in Patients With Advanced Hepatocellular Carcinoma.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/00223
Record Dates: First submitted 2021-08-31; First posted 2021-10-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: MTL-CEBPA; Atezolizumab; Bevacizumab
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Advanced HCC patients (Experimental): Patients will receive treatment as outlined until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, and clinical status. If scheduled dosing and study assessments are precluded because of a holiday, weekend, or other event, then dosing may be postponed to the soonest following date, with subsequent dosing continuing on a 21-day schedule. If treatment was postponed for fewer than 3 days, the patient can resume the original schedule.
  Interventions: Drug: MTL-CEBPA; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: MTL-CEBPA — The starting dose will be at dose level 1. For cycle 1 only, there will be a lead-in period whereby patients will receive one dose of MTL-CEBPA, 7 days prior to cycle 1 day 1. MTL-CEBPA is then administered on Day 1 and 8 of each cycle, atezolizumab is administered on Day 1 of each cycle and bevacizumab is administered on Day 1 of each cycle. One cycle of treatment consists of 21 days.
Drug: Atezolizumab — The starting dose will be at dose level 1. For cycle 1 only, there will be a lead-in period whereby patients will receive one dose of MTL-CEBPA, 7 days prior to cycle 1 day 1. MTL-CEBPA is then administered on Day 1 and 8 of each cycle, atezolizumab is administered on Day 1 of each cycle and bevacizumab is administered on Day 1 of each cycle. One cycle of treatment consists of 21 days.
Drug: Bevacizumab — The starting dose will be at dose level 1. For cycle 1 only, there will be a lead-in period whereby patients will receive one dose of MTL-CEBPA, 7 days prior to cycle 1 day 1. MTL-CEBPA is then administered on Day 1 and 8 of each cycle, atezolizumab is administered on Day 1 of each cycle and bevacizumab is administered on Day 1 of each cycle. One cycle of treatment consists of 21 days.

SUMMARY:
This is a single-center, phase 1, open label, dose-escalation study of MTL-CEBPA co-administered with atezolizumab and bevacizumab to assess the PK, PD, and potential toxicities of the drug combination in advanced HCC patients, and to determine the MTD, OBD or RP2D. The sample size employed is a minimally modified standard 3+3 cohort model commonly used in Phase I oncology studies. Once determined, the MTD/OBD/RP2D will be administered to an Expansion Cohort (Phase Ib) of 10 additional patients with advanced HCC.

DETAILED DESCRIPTION:
Objectives and Study Endpoints

Study Objectives

1. Primary Objectives

   * To determine the safety and tolerability of combination treatment MTL-CEBPA + atezolizumab + bevacizumab and determine the maximum tolerated dose (MTD) or optimum biologic dose (OBD), dose-limiting toxicities (DLTs), and recommended phase 2 dose (RP2D) for patients with advanced HCC.
   * To determine the anti-tumor response using RECIST v1.1. of combination treatment MTL-CEBPA + atezolizumab + bevacizumab.
2. Secondary Objectives

   * To assess the pharmacodynamics (PD) of combination treatment MTL-CEBPA + atezolizumab + bevacizumab notably on the effects on TIME (tumor immune microenvironment).
   * To assess the pharmacokinetics (PK) of combination treatment MTL-CEBPA + atezolizumab + bevacizumab.
   * To evaluate anti-tumour response using HCC modified RECIST (HCC mRECIST) and immune-modified RECIST (imRECIST) for combination treatment MTL-CEBPA + atezolizumab + bevacizumab in patients with advanced HCC.

Study Endpoints

1. Primary Endpoint

   * Dose escalation part of the study (Phase 1a): the primary endpoint will be dose limiting toxicity (DLT) as defined in Section 4.4.2.
   * Dose expansion part of the study (Phase 1b): the primary endpoint will be objective response rate (ORR) using RECIST v1.1 for a response duration of at least 6 weeks.
2. Secondary Endpoints

   In phase 1a and 1b, the secondary endpoints are:
   * The frequency of adverse events graded according to toxicity criteria (CTCAE v5.0) and categorized by body system and diagnosis.
   * PK parameters defined by the maximum plasma concentration (Cmax), time to maximum plasma concentration (Tmax), area under the plasma concentration curve (AUC) and the half-life of MTL-CEBPA after intravenous administration.
   * Evaluation of changes in surrogate biomarkers, notably changes in levels of MDSCs

   In phase 1b, additional secondary endpoints include:
   * Progression free survival (PFS) defined as time from first dose of study drug to until progression or relapse, or death from any cause, whichever occurred first
   * Overall survival (OS) defined as time from first dose of study drug until death from any cause.
3. Exploratory Endpoints

In phase 1a and 1b, exploratory endpoints are:

* Objective response rate (ORR) using HCC mRECIST and imRECIST.
* Changes from baseline of protein expression levels in blood and tumour tissue (including CEBPα and P21) as well as mRNA expression levels in blood (including CEBPA mRNA) will be evaluated.
* Changes in Tumour Mutational Burden (TMB) and PD-L1 status (biopsy samples) will both be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet ALL of the following inclusion criteria to participate in this study:

  * Signed informed consent.
  * Age ≥ 21 years
  * Life expectancy >3 months
  * Eastern Cooperative Oncology Group (ECOG) performance status (ECOG PS) score of 0 or 1
  * Histologically confirmed metastatic and/or unresectable HCC with cirrhosis resulting from hepatitis B, hepatitis C, alcohol-related liver disease or any other aetiology OR Histologically confirmed metastatic and/or unresectable HCC with or without cirrhosis
  * Child-Pugh class A
  * Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies
  * No prior systemic therapy (including systemic investigational agents) for HCC
  * At least one measurable (per RECIST v1.1) untreated lesion
  * Patients who received prior local therapy (e.g., radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial embolization, etc.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST version 1.1.
  * Acceptable laboratory parameters, as demonstrated by:

    1. Platelets ≥ 75 x 109/L
    2. Serum albumin ≥ 28 g/L
    3. ALT and AST ≤ 5 x ULN
    4. Bilirubin ≤ 3 x ULN
    5. Absolute neutrophil count ≥ 1.5 x 109/L
    6. Haemoglobin ≥ 9.0 g/dL. Patients may be transfused to meet this criterion.
    7. INR < 1.7 (for patients not receiving therapeutic anticoagulation)
    8. Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
    9. Urine dipstick for proteinuria < 2+. Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 2 g of protein in 24 hours.
  * For patients with active hepatitis B virus (HBV): HBV DNA < 500 IU/mL obtained within 28 days prior to initiation of study treatment, and on anti-HBV treatment (per local standard of care; e.g., entecavir) prior to study entry and willingness to continue treatment for the length of the study
  * By signing the consent form patients will confirm they agree to undergo all mandated biopsies, if this can be performed safely. Waiver of biopsy may be granted on a case-to-case basis after discussion with the PI.
  * Willingness and ability to comply with all protocol requirements including scheduled visits, treatment plans, laboratory tests and other study procedures
  * Women of childbearing potential (WOCBP) must have a negative pregnancy test at study entry. Subjects not considered WOCBP are those without menses for ≥ 12 consecutive months, and those who have undergone hysterectomy and/or bilateral salpingo-oophorectomy. WOCBP must be willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study and 6 months after the last dose of treatment.
  * Male participants with partners of child bearing potential are required to use barrier contraception in addition to having their partner use another method of contraception during the study and for 6 months after the last dose of treatment. Male participants will also be advised to abstain from sexual intercourse with pregnant or lactating women, or to use condoms.
  * Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrolment. Patients who have undergone an EGD within 6 months of prior to initiation of study treatment do not need to repeat the procedure.

Exclusion Criteria:

* Patients should not enter the study if ANY of the following exclusion criteria are fulfilled:

  * Child-Pugh class B or C
  * Patients who have been treated with loco-regional therapy within the last 28 days prior to study treatment initiation
  * Major surgery within the last 28 days prior to study treatment initiation
  * Any systemic therapy or investigational agent in the advanced setting within 28 days prior to initiation of study treatment
  * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies or treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
  * Grade > 1 prior treatment-related toxicity (excluding alopecia) at the time of screening
  * Use of filgrastim or peg-filgrastim 14 days prior to study entry
  * Patients with clinically significant cancer ascites
  * Any episode of bleeding from oesophageal varices or other uncontrolled bleeding within the last 6 months prior to study treatment initiation
  * Patients administered with serum albumin within the last 7 days prior to the first study drug administration
  * Known infection with human immunodeficiency virus (HIV)
  * Known active tuberculosis (TB)
  * Leptomeningeal metastasis
  * Symptomatic brain metastases. Asymptomatic patients with treated brain metastases are eligible, provided that all of the following criteria are met:

    1. Measurable disease, per RECIST v1.1, must be present outside the CNS.
    2. The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
    3. There is no evidence of interim progression between completion of CNS-directed therapy and initiation of study treatment.
    4. The patient has not undergone stereotactic, whole-brain radiotherapy, and/or neurosurgical resection within 28 days prior to initiation of study treatment.
    5. Are not receiving corticosteroids or corticosteroids in doses no greater than physiological replacement (e.g., dexamethasone < 1.5 mg/day). Anticonvulsant therapy at a stable dose is permitted.
    6. Asymptomatic patients with brain metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.
  * Treatment with strong CYP3A4 inducers within 14 days prior to initiation of study treatment, including rifampin (and its analogues) or St. John's wort.
  * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

Patients who received acute, low-dose (≤10 mg prednisolone or equivalent per day), systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy, premedication to prevent infusion reaction) are eligible for the study after PI approval has been obtained. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

* Inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg. Anti-hypertensive therapy to achieve these parameters is allowed.
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment
* History of significant hemoptysis (≥2.5 mL of bright red blood per episode) within 1 month prior to initiation of study treatment
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Patients on anticoagulation for therapeutic purposes and is unable to discontinue anti-coagulation (see section 4.12.3 for prohibited anti-coagulant drugs)
* Patients on warfarin (for therapeutic or prophylactic purpose)
* History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, bowel obstruction or intra-abdominal abscess within 6 months prior to initiation of study treatment.
* Clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding prior to initiation of study treatment. Patients with signs/symptoms of sub-/occlusive syndrome/intestinal obstruction at time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for symptom resolution.
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
* Radiotherapy within 28 days prior to initiation of study treatment, except palliative radiotherapy to bone lesions within 7 days prior to initiation of study treatment.
* Local therapy to liver (e.g., radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial embolization, etc.) within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  2. Patients with vitiligo or alopecia
  3. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  4. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided that they do not require systemic therapy
  5. Patients with celiac disease controlled by diet alone.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* History of congenital long QT syndrome or corrected QT interval > and = 500 ms (calculated with use of the Fridericia method) at screening.
* Signs and symptoms of heart failure characterised as greater than the New York Heart Association (NYHA) Class I or other clinically significant cardiac abnormalities (including history of myocardial infarction) including stable abnormalities.
* Patients with history of stem cell / solid organ transplantation.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Pregnant or lactating women
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the last dose of atezolizumab.
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Any other condition (e.g., known or suspected poor compliance, etc.) that, in the judgment of the investigator, may affect the participant's ability to follow the protocol specific procedures.
* Known hypersensitivity to Chinese hamster ovary cell products or the active substance (MTL-CEBPA, atezolizumab or bevacizumab).
* History of malignancy other than HCC within 5 years prior to screening, with the exception of adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding.
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evaluable for Objective Response | 5 years
  Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response (using RECIST v1.1)
Evaluable Non-Target Disease Response | 5 years
  Patients who have lesions present at baseline that are evaluable but do not meet the definitions of measurable disease, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for non-target lesion assessment. The response assessment is based on the presence, absence, or unequivocal progression of the lesions.

SECONDARY OUTCOMES:
Measurable Disease | 5 years
  Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by chest x-ray, as ≥ 10 mm with CT scan, or ≥ 10 mm with calipers by clinical exam. All tumor measurements must be recorded in millimeters.
Evaluation of Best Overall Response | 5 years
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence or non-protocol therapy (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ean Chee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078